CLINICAL TRIAL: NCT07341061
Title: Comprehensive Geriatric Assessment in Primary Care for Older Adults Across Levels of Frailty
Brief Title: Comprehensive Geriatric Assessment in Primary Care
Acronym: PC-CGA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Barry Clarke, Principle Investigator, Nova Scotia Health Authority
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 1032253; 2021-1962 (Other Grant/Funding Number: Research Nova Scotia)
Record Dates: First submitted 2025-12-17; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Frailty; Aging; Geriatric Syndromes; Mobility Limitation; Functional Decline; Sedentary Lifestyle
Keywords: Frailty; eCGA; electronic Comprehensive Geriatric Assessment; Primary Care; Frailty Index; Clinical Frailty Scale; Older Adults; Healthy Aging; Physical Activity Intervention; Exercise Intervention; Geriatric Assessment
MeSH Terms: conditions — Frailty; Mobility Limitation; Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: Randomized, delayed-start, parallel design comparing immediate versus delayed personalized physical activity intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group AB - immediate exercise group (Experimental): Participants begin the Personalized Approach for Healthy Aging (PAHA) physical activity intervention immediately after basline assessment. The intervention includes individualized goal setting using Goal Attainment Scaling, tailored exercise prescription, and structured follow-up contacts with a Clinical Exercise Physiologist.
  Interventions: Behavioral: Personalized Approach for Healthy Aging (PAHA)
- Group BA - 6-month delayed exercise group (Active Comparator): Participants begin the PAHA physical activity intervention after a delayed-start period. They complete the same assessments and receive the same individualized exercise program as Group AB (immediately exercise group) but begin the intervention later in the study.
  Interventions: Behavioral: Personalized Approach for Healthy Aging (PAHA)

INTERVENTIONS:
Behavioral: Personalized Approach for Healthy Aging (PAHA) — A personalized physical activity and behaviour-change program delivered by a Clinical Exercise Physiologist, including individualized goal setting, tailored home-based exercise prescriptions, and structured follow-up contacts (telephone or virtual) over 6 months.

SUMMARY:
This study evaluates the feasibility and acceptability of implementing the electronic Comprehensive Geriatric Assessment (eCGA) in primary care for adults aged 65 years and older. The study examines how frailty changes over 12 months, how patient self-assessments compare with physician assessments, and how patients perceive the value of the eCGA when used as part of routine care.

The study also includes an interventional randomized sub-study (PAHA), in which eligible participants receive a personalized physical activity program developed by a Clinical Exercise Physiologist. Participants are randomized to either an immediate-start or delayed-start exercise group, allowing assessment of the effects of a tailored activity intervention on frailty, physical activity participation, and goal attainment.

Findings will inform how eCGA tools and personalized activity interventions can be integrated into primary care to support healthy aging and frailty management.

DETAILED DESCRIPTION:
This study investigates the use of the electronic Comprehensive Geriatric Assessment (eCGA) in primary care as a structured approach to identifying frailty, monitoring change over time, and informing individualized care planning for older adults. The eCGA is an electronic adaptation of the Comprehensive Geriatric Assessment used in geriatric care, integrated into the TELUS electronic medical record used in Nova Scotia. Embedding the eCGA directly within the EMR is designed to improve feasibility and uptake by allowing primary care physicians to efficiently review key domains of mobility, cognition, mood, comorbidities, medications, and daily function during routine care encounters to generate a frailty index (FI).

The main study is a prospective, longitudinal cohort conducted in a primary care clinic. Up to 120 adults aged 65 and older will complete baseline eCGA assessments, patient-reported frailty and health questionnaires with follow-up at 12-months. We will investigate changes in frailty status, concordance between physician and patient frailty assessments (eCGA Frailty Index, Clinical Frailty Scale, Pictorial Fit-to-Frail Scale, Health Questionnaire - Frailty Index), patient experiences with the eCGA process, and health service utilization. Quantitative analyses include descriptive statistics, paired comparisons, one-way ANOVA models, correlation analyses, and regression models to identify predictors of frailty change. Qualitative semi-structured interviews will explore participants' perspectives on the acceptability and perceived clinical value of the eCGA.

The study also includes a randomized interventional sub-study-the Personalized Approach for Healthy Aging (PAHA). Sixty to 120 participants will be randomized into two groups.

Group AB (Immediate Exercise Group) will receive a tailored physical activity intervention beginning at baseline.

Group BA (Delayed Exercise Group) will receive the same intervention beginning after an initial waiting period.

The intervention is delivered by a Clinical Exercise Physiologist and includes individualized goal setting using Goal Attainment Scaling, a tailored exercise prescription, and structured follow-up contacts (weekly in month 1, biweekly in month 2, then monthly to month 6. This will vary by participant as needed). Randomization is stratified by Clinical Frailty Scale score.

The PAHA sub-study evaluates whether a personalized exercise intervention can improve physical activity levels (Physical Activity Scale for the Elderly), frailty progression, and individualized goals. Mixed-effects models will be used to examine longitudinal changes in activity and frailty, with "time zero" defined as the start of the intervention for each participant. Time points prior to and after the start of the intervention will be analyzed to evaluate treatment effects, carry-over effects, and sequence effects. Participants who withdraw early will still contribute available data, consistent with mixed-model analytic methods.

Safety monitoring is integrated into both clinical practice and the study design. All participants undergo a physician assessment prior to sub-study enrollment; referrals to physiotherapy or occupational therapy occur when clinically appropriate. The Clinical Exercise Physiologist monitors symptoms, adherence, and adverse events at each contact and modifies exercise prescriptions as necessary. All serious adverse events potentially related to the intervention are reviewed by the Principal Investigator and reported in accordance with institutional policy.

Qualitative and quantitative data will be triangulated to provide a comprehensive understanding of the feasibility, acceptability, and potential clinical impact of integrating frailty assessment and tailored physical activity support into routine primary care for older adults.

ELIGIBILITY:
Inclusion Criteria:

* Older adult patients receiving care at the Dalhousie Family Medicine Clinic and scheduled to undergo an eCGA as part of routine primary care.
* Fluent in English and able to respond to interview and questionnaire items.
* Able to provide informed consent; or, if judged unable to consent, able to provide assent AND has a substitute decision maker (SDM) who is willing to provide informed consent on their behalf.
* (PAHA sub-study) Enrolled in the main eCGA study, willing to participate in a personalized physical activity- program, and available for follow-up contact.

Exclusion Criteria:

* Not scheduled for, or not receiving, an eCGA at the investigator's family medicine clinic.
* Unable to communicate in English, such that questionnaires and interviews cannot be completed.
* Unable to provide informed consent and no SDM available or willing to consent on the patient's behalf.
* (PAHA sub-study) Deemed unsuitable for the physical activity intervention by the treating family physician (e.g., medical or functional condition that, in the physician's judgment, makes participation in light-moderate exercise unsafe).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01-12 (Estimated); Primary Completion 2027-07-12 (Estimated); Study Completion 2029-01-12 (Estimated)

PRIMARY OUTCOMES:
Comprehensive Geriatric Assessment - Frailty Index | Assessed at baseline and at 12-month follow-up.
  A comprehensive geriatric assessment (CGA) of the participants' global health state, including their current and relevant past illnesses, medications, cognition, emotion, motivation, health attitude, communication, sleep, pain, control of life, strength, balance, mobility, activities and instrumental activities of daily living, quality of life, lifestyle, and social engagement are assessed. Information to inform the CGA is derived from participant interviews, structured assessments and tests, and medical record review. Each CGA item will be recoded to a scale from 0 to 1, with 0 representing no deficit and 1 representing the full deficit. The total Frailty Index score will be calculated by dividing the sum of the variables' recoded values (the sum of the deficits) by the number of variables measured for that person. The range of the frailty index score is between 0 and 1, where higher scores indicate greater frailty.
Health Questionnaire - Frailty Index | Baseline and 12-month follow-up.
  The health questionnaire includes questions related to self-rated health, chronic conditions, activities of daily living, instrumental activities of daily living, cognitive function, and mental health. Responses to each question will be coded on a scale from 0 to 1, with 0 representing no deficit and 1 representing the full deficit. The total health questionnaire Frailty Index score will be calculated by dividing the sum of the variables' coded values (the sum of the deficits) by the number of variables measured for that person. The range of the frailty index score is between 0 and 1, where higher scores indicate greater frailty.
Clinical Frailty Scale | Baseline and 12-month follow-up
  The Clinical Frailty Scale (CFS) broadly stratifies degrees of fitness and frailty on a 9-point scale where higher scores indicate greater risk: 1-very fit; 2-fit; 3-managing well; 4-living with very mild frailty; 5- living with mild frailty; 6-living with moderate frailty; 7-living with severe frailty; 8- living with very severe frailty; and 9-terminally ill. The score is based on clinical judgment as part of the comprehensive geriatric assessment.
Pictorial Fit-Frail Scale | Baseline and 12-month follow-up.
  This is a brief, picture-based frailty assessment designed so patients, caregivers, or clinicians can rate current health status common across 14 domains (e.g., mobility, function, cognition, mood, nutrition, comorbidity) using simple visual panels. This scale will be completed separately by participants (self-administered version) and health care professionals (PFFS-HCP). For each domain, the level representing least or no impairment (first picture on the left) is scored 0, the next level (second picture from the left) as 1, etc. The minimum score for each domain is 0; the maximum score for each domain ranges from 2 to 5. Total Pictorial Fit-Frail Scale scores are calculated by summing the scores across domains. The final summed score ranges from 0 (no frailty; very fit) to 43 (severely frail).
Physical Activity Scale for the Elderly | Group AB: Baseline, 3 months, 6 months, and 12 months Group BA: Baseline, 6 months, 9 months, and 12 months.
  The Physical Activity Scale for the Elderly (PASE) quantifies the frequency, duration, and intensity of physical activities, and sedentary time. The scale includes 10 questions that collect information about physical activities performed over the past week, including leisure activities, household activities, work, and volunteering (e.g., walking, caring for another person).
  The responses for each activity are used to calculate a total score. Scores range from 0 to over 400, with higher scores representing greater activity levels. The Physical Activity Scale for the Elderly will be administered by the Clinical Exercise Physiologist. It will only be administered to participants who consent to participate in the sub-study.
Patient acceptability of eCGA | Baseline with follow-up at 12-months.
  Acceptability of the electronic Comprehensive Geriatric Assessment (eCGA) as reported by participants using an 18-item survey administered post-CGA to assess ease of completion, understanding, perceived usefulness, and overall satisfaction. Each item is scored on a 5-point Likert scale where 1 indicates strong agreement and 5 indicates strong disagreement. The acceptability score will be calculated by summing all item scores. The total score will range from 18 (best outcome) to 90 (worst outcome).

SECONDARY OUTCOMES:
Goal Attainment (PAHA Sub-Study) | Group AB: Baseline with follow-up at 3-, 6-, and 12-months. Group BA: Baseline with follow-up at 6-, 9-, and 12-months.
  Goals are constructed on a 5-point scale ranging from +2 (much better than the expected outcome) to -2 (much worse than the expected outcome), where the participant's baseline status is set as -1 and the expected outcome (i.e., desired goal) is set as 0. Goals are set at baseline with the Clinical Exercise Physiologist who reviews attainment status with participants at each follow-up. Mean Goal Attainment scores and proportion of goals achieved will be reported. Goal Attainment Scaling is individualized in that participants select goal that are personally relevant. Summarizing this individualized information is accomplished using a formula that accounts for the number of goals set and variations in attainment (total score range 17 - 82 with higher scores indicating greater goal achievement).
Qualitative experience of the eCGA and PAHA | Interviews conducted approximately 12 months after baseline.
  Semi-structured interviews at 12 months will explore participants' experiences of the eCGA process and, for PAHA participants, the personalized exercise program (acceptability, feasibility, perceived benefits, and barriers). Transcripts will be analyzed using thematic analysis to identify key themes informing implementation.
Number of falls and fractures | At 12-month follow-up.
  Falls and fractures within the past year will be self-reported.
Transition to institution or higher level of care | At 12-month follow-up
  Number of participants who changed their living arrangement during the study period (12-months), including transition to institution or higher level of care (e.g. from community to assisted living or from assisted living to nursing home)
Hospital and Emergency Department admissions | At 12-month follow-up
  Counts and length of emergency department visits and hospital admissions per participant during the study period (12-months), obtained from patient report and chart review.
Number of deaths | At 12-month follow-up
  Count of participants who died before their 12-month follow-up would have occurred.

CONTACTS AND LOCATIONS:
Overall Officials: Barry Clarke, MD, Principal Investigator — Nova Scotia Health

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to institutional privacy policies and the terms of participant consent. Summary results will be made available through publications and ClinicalTrials.gov.